CLINICAL TRIAL: NCT02542059
Title: Visualizing Beta Cells in Patients With Remission of T2DM After Bariatric Surgery
Brief Title: Visualizing Beta Cells After Bariatric Surgery
Acronym: GLP1-bar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL51058.091.14
Record Dates: First submitted 2015-08-18; First posted 2015-09-04 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Responders: Patients with resolved type 2 diabetes after bariatric surgery, will undergo 68Ga-exendin PET/CT
  Interventions: Radiation: 68Ga-exendin PET/CT
- Non-responders: Patients with unresolved type 2 diabetes after bariatric surgery, will undergo 68Ga-exendin PET/CT
  Interventions: Radiation: 68Ga-exendin PET/CT

INTERVENTIONS:
Radiation: 68Ga-exendin PET/CT — 68Ga-exendin PET/CT
  Other Names: GLP-1 receptor PET/CT

SUMMARY:
In order to evaluate the difference in beta cell mass in patients with and without complete resolution of type 2 diabetes mellitus (T2DM) after Roux en Y gastric bypass (RYGB) investigators aim to compare quantitative PET imaging of the pancreas between these patient groups.

These highly relevant data will provide investigators with more information on the possible role of beta cell mass in the mechanisms behind resolution of T2DM after bariatric surgery. This would be of great interest for the assessment of RYGB as an alternative therapy in patients with T2DM with a BMI <35, who currently do not meet the international guidelines for bariatric surgery.

DETAILED DESCRIPTION:
Obesity and T2DM The prevalence of Type 2 Diabetes Mellitus (T2D) in the Netherlands is 600.000-800.000 and each year ~70.000 new patients are diagnosed. This increasing number of patients with T2D is closely correlated with the obesity epidemic. In women, over 50% of T2D risk can be accounted for by obesity. Also, over 85% of T2D patients are overweight and ~50% are obese.

Obese patients with T2D not only have elevated glucose levels but are also at risk to develop dyslipidemia and hypertension. This clustering of cardiovascular risk factors leads to an increased risk of micro-and macrovascular long-term complications. In fact, patients with T2D have a 2-4 times increased risk for cardiovascular disease. These complications seriously decrease the quality of life and life expectancy of T2D patients. The burden of this disease not only affects these patients but our society as well. Health care costs with respect to diabetes amounted 814 million euro in 2005 in the Netherlands and indirect costs because of absence of work are unknown but thought to be substantial.

Weight loss is perhaps the most important therapeutic intervention in obese patients with T2D. Weight loss intervenes in the underlying pathophysiology and restores insulin sensitivity and sometimes even insulin secretion. In addition, it improves dyslipidemia and hypertension. In contrast, most pharmacological interventions only relieve the symptoms of the complex disease process underlying T2DM whilst the disease process itself is not addressed and even progresses in the course of time. Unfortunately, the effect of weight loss interventions such as diet and lifestyle or even drugs is often modest (3-5 kg) and short-lived.

Bariatric surgery and T2DM remission Weight reducing surgery, i.e. bariatric surgery, is the only intervention that leads to persistent weight loss and it is superior above conventional (non-surgical) treatment.

Bariatric surgery can be divided into restrictive (gastric band) and malabsorptive procedures (biliopancreatic diversion) or a combination of the 2 (Roux-en-Y Gastric Bypass, RYGB).

The current indications are BMI > 40 kg/m2 or BMI > 35 kg/m2 with co-morbidities like T2D. The greater the malabsorptive component, the greater the effect on weight loss.

Meta-analyses also showed spectacular metabolic improvement of bariatric surgery in obese patients with T2D.

The mechanism of diabetes resolution after RYGB is not completely understood and there is evidence that it might not be completely dependent on weight loss. While significant weight loss has not yet been achieved within days after the surgery, glycemic control has been found to occur already at this time. Also, the improvement in glucose control after gastric bypass is greater than with equivalent weight loss obtained by dietary intervention or purely restrictive bariatric procedures. There are several hypotheses concerning the weight-independent effects of bariatric surgery on insulin secretion. The most popular ones are the 'hindgut-hypothesis', which states that expedited delivery of nutrients to the distal intestine enhances the secretion of intestinal peptides like glucagon-like-peptide 1 (GLP1) and peptide YY and the 'foregut hypothesis', which states that the exclusion of the duodenum and proximal jejunum from the transit of nutrients results in changes in secretion of intestinal peptides. However, several other mechanisms, both in- and outside the intestines might play a role.

While improvement of beta cell function has been reported in both healthy individuals as well as T2D patients after RYGB it is unclear whether the actual beta cell mass is subject to change after bariatric surgery. In Goto-Kakizaki rats duodenal jejunal bypass was found to increase pancreatic concentrations of vesicular monoamine transporter type 2 (VMAT2), a biomarker for beta cells. Furthermore, an increase in beta cell mass, beta cell number and extra islet beta cells was found after RYGB in a porcine model. However, there are only few studies in humans, with conflicting results.

The benefit of bariatric surgery on glycemic control in morbidly obese patients (BMI 35 kg/m2 or more) with T2DM is confirmed and has been accepted as an alternative therapy in this patient population for treatment of T2DM by the Diabetes Surgery Summit Consensus Conference (DSS), which was participated by 50 experts and endorsed by multiple international scientific societies (such as American Diabetes Association (ADA) and the International Federation for the Surgery of Obesity and Metabolic diseases (IFSO)) and the International Diabetes Federation Taskforce on epidemioloy and Prevention of Diabetes, a consensus working group of diabetologists, surgeons and public health experts. They also consider expanding the indications for bariatric surgery in obese patients with T2D who currently don't meet the international guidelines for bariatric surgery. In this regard, more information on the effects of bariatric surgery on beta cell function and beta cell mass would be helpful. If this information could be obtained preoperatively this would improve the selection of patients who would benefit from bariatric surgery.

Imaging of beta cells in vivo Reliable, sensitive and specific visualization of living pancreatic beta cells in vivo is important to broaden our understanding of resolution of T2D after bariatric surgery. Reliable quantification of the remaining beta cell mass will lead to a better assessment of beta cell function after bariatric surgery. This could lead to a better understanding of the relative importance of factors leading to the recovery of glycemic control. This could help in the consideration whether to expand the indications for bariatric surgery to patients with T2D who currently do not meet the criteria (BMI<35).

ELIGIBILITY:
Inclusion Criteria:

For responders:

* Obese T2D patient who had undergone RYGB at least 1 year earlier
* Signed informed consent
* Complete resolution of T2D after surgery

For non-responders:

* Obese T2D patient who had undergone RYGB at least 1 year earlier
* Signed informed consent
* No complete resolution of T2D after surgery

Exclusion Criteria:

* Previous treatment with synthetic exendin
* Breast feeding
* Pregnancy or the wish to become pregnant within 6 months
* renal dysfunction
* Age < 18 years
* Incapacitated
* No signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Indiciduals who have undergone RYGB at least 1 year earlier at the Rijnstate Hospital in Arnhem.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2015-08; Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Beta cell mass measured by uptake of 68Ga-exendin in the pancreas on PET images | 1 year

SECONDARY OUTCOMES:
Comparing uptake of 68Ga-exendin in the pancreas with blood glucose and insulin measured after glucose ingestion and arginine infusion | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gotthardt, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem, Gelderland
  - RadboudUMC, Nijmegen, Gelderland

REFERENCES:
- [Derived] Tokgoz S, Deden LN, Hofboer A, Meijer RI, Hazebroek EJ, van Bon AC, de Galan BE, Tack CJ, Boss M, Gotthardt M. Beta cell function and mass in individuals with and without remission of type 2 diabetes after Roux-en-Y gastric bypass. Diabetologia. 2026 Jan 20. doi: 10.1007/s00125-025-06659-1. Online ahead of print. PMID 41555052